CLINICAL TRIAL: NCT05726825
Title: Randomized, Prospective, Multicenter, Open-label, Controlled, Parallel-group Trial Investigating the Efficacy of Add-on Plasma Exchange As an Adjunctive Strategy Against Septic Shock - 2
Brief Title: Efficacy of Add-on Plasma Exchange As an Adjunctive Strategy Against Septic Shock
Acronym: EXCHANGE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXCHANGE-2
Record Dates: First submitted 2023-01-16; First posted 2023-02-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: Septic Shock; Sepsis; Multi-organ failure; Extracorporeal therapy; Plasmapheresis
MeSH Terms: conditions — Shock, Septic; Sepsis; Multiple Organ Failure | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Plasma Exchange (TPE) (Experimental): 1 x TPE with donor Fresh Frozen Plasma (FFPs) (1.2 x individual plasma volume) within the first 6 hrs after randomization.
  A second TPE can be performed if the patient remains vasopressor dependent ≥ 0.4 ug/kg/min within 24 hours after the first intervention.
  Interventions: Device: Therapeutic Plasma Exchange (TPE)
- Standard of Care (SOC) (No Intervention): Non-interventional standard of care

INTERVENTIONS:
Device: Therapeutic Plasma Exchange (TPE) — The TPE treatment will be initiated within 6 hrs after randomization. Duration of TPE treatment is approximately 120-180 minutes. An additional second TPE can be performed if the patient remains vasopressor dependent ≥ 0.4 ug/kg/min after 24 hours following the first TPE procedure.
  Both unfractionated heparin (UFH) and citrate may be used as anticoagulant medication.
  To ensure treatment comparability between different patients, we will replace plasma in a fixed ratio of 1.2 x the individual patient's total plasma fluid.
  Arms: Therapeutic Plasma Exchange (TPE)

SUMMARY:
Randomized, prospective, multicenter, open-label, controlled, parallel-group interventional trial to test the adjunctive effect of therapeutic plasma exchange in patients with early septic shock.

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening organ dysfunction caused by a dysregulated host response to an infection; in septic shock profound circulatory, cellular and metabolic abnormalities are associated with an even higher mortality. Sepsis is a major healthcare problem, affecting millions of individuals around the world each year. Its incidence appears to be rising, and the mortality caused by septic shock in Germany in 2015 remains extraordinarily high (58.8%). It is well known - from the pathophysiological point of view - that these patients do not die from their infection per se but rather from multiple organ failure caused by their own overwhelming host response. This fact is so fundamental that it has been implemented as a key part of the 2016 sepsis definition (SEPSIS-3). Despite tremendous efforts during the last decades, innovative approaches targeting this fundamental hallmark of the disease, thereby reducing organ dysfunction, are lacking. Undoubtedly, there is an unmet need to expand the current standard of care for these patients by a more specific intervention.

The investigators hypothesize that early Therapeutic Plasma Exchange (TPE) in the most severely ill individuals will dampen the injurious maladaptive host response by removing injurious mediators thereby limiting organ dysfunction. The potential impact of this trial is of immense clinical relevance as it evaluates a promising adjunctive treatment option for a patient cohort suffering from an extraordinary high mortality. A positive trial result could truly change the current standard of care (SOC) - that is mostly supportive - of septic shock patients. Of note, there is neither a patent nor a direct commercial interest in such a trial.

ELIGIBILITY:
Inclusion Criteria:

* New onset of septic shock (< 24 hrs), (SEPSIS-3 definition)
* Norepinephrine (NE) dose ≥ 0.4 μg/kg/min ≥ 30 min OR NE ≥ 0.3 μg/kg/min + vasopressin (any dose)
* Established vascular access suitable for plasma exchange independent of study inclusion (due to established indication of RRT, expected need for RRT within the next 48 hours or other medical reasons as assessed by treating physician team)

Exclusion Criteria:

* Age < 18 or > 80 years
* Urogenital focus of infection
* Pregnancy
* Heparin-induced thrombocytopenia
* Known reaction against fresh frozen plasma (FFP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | from randomization up to 28 days following randomization

SECONDARY OUTCOMES:
Mean daily Sequential Organ Failure Score (SOFA) score over the first 7 days (KEY secondary outcome) | from randomization up to 7 days following randomization
  Per-patient mean daily SOFA score over the first 7 days, ranging from 0-24 points with higher scores indicating more severe organ dysfunction
Organ support free days until day 28 (KEY secondary outcome) | from randomization up to 28 days following randomization
  total days free of invasive ventilation, vasopressors/inotrops and renal replacement therapy (RRT) until day 28
90-day mortality | from randomization up to 90 days following randomization
Intensive Care unit (ICU) length of stay | from randomization until ICU discharge
  total days in ICU
Hospital length of stay | from randomization until hospital discharge
  total days in hospital
Basic Hemodynamics | at days 1-7 following randomization
  includes: Norepinephrine- [µg/kg/min], Dobutamine [µg/kg/min], Epinephrine- [µg/kg/min] and Vasopressin-dose [U/kg/min], Vasocative-inotropic (VIS) Score with higher scores indicating higher vasopressor/inotropic support, Mean arterial pressure (MAP, [mmHg]), Heart Rate (HR, [1/min]), Central venous pressure (CVP, [mmHg]) and Central-Venous Oxygen Saturation (ScvO2, [%]) at 0 and 12 hrs, d1-7
Extended Hemodynamics | at days 1-7 following randomization
  includes: Cardiac Index (CI, [l/min/m2]), Global End-Diastolic Volume Index (GEDI, [ml/m2]), Sytemic Vascular Resistance Index (SVRI, [dyn*s*cm-5*m2]), Stroke Volume Variation (SVV, [%] ), Extravascular Lung Water Index (ELWI, [ml/kg]) and Pulmonar Vascular Permeability Index (PVPI) at at 0 and 12 hrs, d1-7
Arterial blood gas analysis | at days 1-7 following randomization
  includes: pH, PCO2 [mmHg], HCO3- [mmol], PO2 [mmHg], Lactate [mmol/l] at 0 and 12 hrs, d1-7
Respiratory function | at days 1-7 following randomization
  includes: pO2/FiO2, Tidal Volume (VT, [ml]), Positive End-Exspiratory Pressure (PEEP, [cmH2O]), Peak-Pressure (Ppeak, [cmH2O]), Plateau-Pressure (Pplat, [cmH2O]), Respiratory Rate (RR, [1/min]), Inspiratory Time (Tinsp, [s]), Inspiratory-Flow and End-tidal-CO2 (etCO2, [mmHg]) at 0 and 12 hrs, d1-7
Renal function | at days 1-7 following randomization and at ICU discharge
  includes: Presence of Acute kindey injury (AKI), AKI stage (KDIGO definition) stage 1-3 with higher stage indicating worse renal function, Need for Renal Replacement Therapy (RRT), Estimated Glomerular Filtration Rate (eGFR following CKD-EPI equation) [ml/min], Fluid intake [ml/d], Urine output [ml/d], Ultrafiltration and Net daily fluid balance [ml/d] at 0 and 12 hrs, d1-7 and at ICU discharge
Liver Function | at days 1-7 following randomization and at ICU discharge
  includes: Bilirubin, Aspartate aminotransferase (AST, [U/l]), Alanine aminotransferase (ALT, [U/l]), Alkaline phosphatase (AP, [U/l]), Gamma-glutamyl transferase (GGT, [U/l]), Cholinesterase (CHE, [kU/l]) and Albumin [g/l] at 0 and 12 hrs, d1-7 and at ICU discharge
Sepsis associated coagulopathy | at days 1-7 following randomization
  includes: Differential blood count including schistocytes [%], Fibrinogen [g/l] , D-Dimer [mg/l], International Normalized Ratio (INR), Lactate dehydrogenase (LDH, [U/l]), Antithrombin-III (AT-III, [%]), Protein C [%] and International Society on Thrombosis and Hemostasis- Disseminated Intravscular Coagulation Score (ISTH-DIC, [U/l]) ranging from 0-8 points with higher values indication more severe DIC at 0 and 12 hrs, d1-7, A disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 (ADAMTS13, [%]) and von-Willebrand-Factor Antigen (vWF:Ag,[IU/l]) at 0 and 24 hrs
Inflammatory response | at days 1-7 following randomization
  includes: C-reactive protein (CRP, [mg/l]), Procalcitonin (PCT, [ug/l]), Interleukin-6 (IL-6, [ng/ml]), Ferritin [ug/l] and Neutrophil/Lymphocyte ratio at 0 and 12 hrs, d1-7
Cardiac function | at days 1-7 following randomization and at ICU discharge
  includes: Creatine kinase (CK, [U/l]), Myoglobin [ug/l], Troponin T [ng/l], NT-proBNP [ng/l] at 0 and 12 hrs, d1-7 and at ICU discharge
Secondary infections | from randomization until hospital discharge
  includes: incidence and type of secondary infections until ICU and hospital discharge, incidence of viral (HSV, EBV, CMV) reactivation at d7 and d14

OTHER OUTCOMES:
Safety Endpoints | from randomization until day 7 following randomization
  includes: Incidence of bleeding, allergic reactions, Transfusion associated lung injury (TRALI), severe thrombocytopenia (< 5000/µl) and (other) severe adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha David, Prof. Dr., Principal Investigator — University of Zurich; Klaus Stahl, PD Dr., Principal Investigator — Hannover Medical School; Christian Bode, PD Dr., Principal Investigator — University Hospital, Bonn
Locations (25):
- Austria (2):
  - University Hospital Innsbruck, Innsbruck
  - University Hospital Vienna, Vienna
- Germany (21):
  - St. Joseph Hospital, Berlin
  - University Hospital Berlin Charite, Berlin
  - University Hospital Bonn, Bonn
  - Hospital Braunschweig, Braunschweig
  - Hospital Bremerhaven, Bremerhaven
  - Hospital Cologne Meerheim, Cologne
  - University Hospital Cologne, Cologne
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Halle, Halle
  - University Hospital Hamburg (UKE), Hamburg
  - Hannover Medical School Anesthesiology, Hanover
  - Hannover Medical School Internal Medicine, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Jena, Jena
  - University Hospital Kiel, Kiel
  - Hospital Magdeburg, Magdeburg
  - University Hospital Munich (TUM) Anesthesiology, Munich
  - University Hospital Munich (TUM) Internal Medicine, Munich
  - University Hospital Muenster Anesthesiology, Münster
  - University Hospital Rostock, Rostock
- Switzerland (2):
  - University Hospital Bern, Bern
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knaup H, Stahl K, Schmidt BMW, Idowu TO, Busch M, Wiesner O, Welte T, Haller H, Kielstein JT, Hoeper MM, David S. Early therapeutic plasma exchange in septic shock: a prospective open-label nonrandomized pilot study focusing on safety, hemodynamics, vascular barrier function, and biologic markers. Crit Care. 2018 Oct 30;22(1):285. doi: 10.1186/s13054-018-2220-9. PMID 30373638
- [Background] Stahl K, Schmidt JJ, Seeliger B, Schmidt BMW, Welte T, Haller H, Hoeper MM, Budde U, Bode C, David S. Effect of therapeutic plasma exchange on endothelial activation and coagulation-related parameters in septic shock. Crit Care. 2020 Mar 2;24(1):71. doi: 10.1186/s13054-020-2799-5. PMID 32122366
- [Background] Stahl K, Bikker R, Seeliger B, Schmidt JJ, Schenk H, Schmidt BMW, Welte T, Haller H, Hoeper MM, Brand K, David S. Effect of Therapeutic Plasma Exchange on Immunoglobulin Deficiency in Early and Severe Septic Shock. J Intensive Care Med. 2021 Dec;36(12):1491-1497. doi: 10.1177/0885066620965169. Epub 2020 Oct 16. PMID 33063613
- [Background] David S, Bode C, Putensen C, Welte T, Stahl K; EXCHANGE study group. Adjuvant therapeutic plasma exchange in septic shock. Intensive Care Med. 2021 Mar;47(3):352-354. doi: 10.1007/s00134-020-06339-1. Epub 2021 Jan 20. No abstract available. PMID 33471132
- [Background] Stahl K, Hillebrand UC, Kiyan Y, Seeliger B, Schmidt JJ, Schenk H, Pape T, Schmidt BMW, Welte T, Hoeper MM, Sauer A, Wygrecka M, Bode C, Wedemeyer H, Haller H, David S. Effects of therapeutic plasma exchange on the endothelial glycocalyx in septic shock. Intensive Care Med Exp. 2021 Nov 24;9(1):57. doi: 10.1186/s40635-021-00417-4. PMID 34817751
- [Background] Stahl K, Wand P, Seeliger B, Wendel-Garcia PD, Schmidt JJ, Schmidt BMW, Sauer A, Lehmann F, Budde U, Busch M, Wiesner O, Welte T, Haller H, Wedemeyer H, Putensen C, Hoeper MM, Bode C, David S. Clinical and biochemical endpoints and predictors of response to plasma exchange in septic shock: results from a randomized controlled trial. Crit Care. 2022 May 12;26(1):134. doi: 10.1186/s13054-022-04003-2. PMID 35551628
- [Derived] David S, Bode C, Stahl K; EXCHANGE-2 Study group. EXCHANGE-2: investigating the efficacy of add-on plasma exchange as an adjunctive strategy against septic shock-a study protocol for a randomized, prospective, multicenter, open-label, controlled, parallel-group trial. Trials. 2023 Apr 15;24(1):277. doi: 10.1186/s13063-023-07300-5. PMID 37061693